CLINICAL TRIAL: NCT00472173
Title: Assessment of a New Apexification Method for Patients Presenting a Non Vital Immature Tooth
Acronym: APEXMTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06236
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Dental Pulp Necrosis
Keywords: Apexification; Pulp necrosis; Calcium hydroxide; MTA; pulp necrosis of an anterior immature tooth
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — mineral trioxide aggregate; Calcium Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium hydroxide (Active Comparator)
  Interventions: Drug: Calcium hydroxide
- MTA (Experimental)
  Interventions: Drug: Mineral Trioxide Aggregate

INTERVENTIONS:
Drug: Mineral Trioxide Aggregate — Apexification treatment of the tooth with Mineral Trioxide Aggregate
  Arms: MTA
Drug: Calcium hydroxide — Apexification treatment of the tooth with Calcium hydroxide
  Arms: Calcium hydroxide

SUMMARY:
Pulp necrosis is one of the main complication of dental trauma. When it happens on an immature tooth, pulp necrosis implies a lack of root maturation and apical closure. A therapy called apexification is required to induce the formation of a calcified apical barrier allowing a permanent and hermetic root filling.The aim of this study is to compare the efficacy of a new apexification method using Mineral Trioxide Aggregate (MTA®) with the reference treatment based on calcium hydroxide repeated stimulations.

DETAILED DESCRIPTION:
36 patients aged 6 to 18 and presenting a non vital immature tooth will be included in the study (inclusion period: 12 months). These patients will be randomly divided into two groups: one treated with MTA®, and the other one with calcium hydroxide. For each patient, the total duration of the study will be 12 months. Recalls will be performed at 15 and 21 days and then at 3, 6 and 12 months to assess by clinical and X-ray exams the main success criterion: presence of a calcified apical barrier or not. Additional criterions such as presence of clinical symptoms or not, apical morphology and depth of this apical barrier will be observed. This randomised prospective therapeutic study will allow to assess the ability of MTA® inducing apexification of a non vital immature tooth. Furthermore, it will be possible to compare for both materials the kinetics of clinical symptoms disappearance and the morphology and depth of apices.

ELIGIBILITY:
Inclusion Criteria:

* Indication of apexification treatment of an anterior immature tooth
* Patients aged 6 to 18
* Enlightened agreement of the patient and his/her legal representatives
* Prerequisite medical examination

Exclusion Criteria:

General disease

* diabetes
* immunosuppression of whatever origin (AIDS, drugs, …)
* severe asthma
* chronical disease requiring treatment
* eating disorders (anorexia, bulimia, malnutrition, …) Oral disease
* periodontal disease
* Administration of corticoids in a period of 3 months preceding the inclusion
* Patient with no social security cover

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Main success criterion: presence of a calcified apical barrier or not at 3, 6 and 12 months | 30 days

SECONDARY OUTCOMES:
Additional criterions :- presence of clinical symptoms or not- apical morphology - depth of this apical barrier At 3, 6 and 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Lasfargues, Dentist PhD, Principal Investigator — Hôpital Bretonneau - Paris; Raphaël SERREAU, MD, PhD, Study Director — URC Paris Centre
Locations (1):
- Hôpital Bretonneau, Paris, France

REFERENCES:
- [Derived] Beslot-Neveu A, Bonte E, Baune B, Serreau R, Aissat F, Quinquis L, Grabar S, Lasfargues JJ. Mineral trioxyde aggregate versus calcium hydroxide in apexification of non vital immature teeth: study protocol for a randomized controlled trial. Trials. 2011 Jul 13;12:174. doi: 10.1186/1745-6215-12-174. PMID 21752247